CLINICAL TRIAL: NCT02075541
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Investigational Vaccine GSK2838504A When Administered to Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GlaxoSmithkline (GSK) Biologicals' Investigational Vaccine GSK2838504A When Administered to Chronic Obstructive Pulmonary Disease (COPD) Patients With Persistent Airflow Obstruction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200157; 2013-003062-13 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Respiratory Disorders
Keywords: Immunogenicity; Observer-blind; Reactogenicity; Chronic Obstructive Pulmonary Disease; Safety
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 10-AS01E group (Experimental): Subjects in this group will receive the investigational NTHi vaccine.
  Interventions: Biological: NTHi-10-AS01E
- Control group (Placebo Comparator): Subjects in this group will receive placebo.
  Interventions: Drug: NaCl Placebo

INTERVENTIONS:
Biological: NTHi-10-AS01E — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: 10-AS01E group
Drug: NaCl Placebo — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Control group

SUMMARY:
The purpose of this Phase II study is to assess the safety, reactogenicity and immunogenicity of the investigational Non-typeable Haemophilus influenzae (NTHi) vaccine in patients with moderate and severe persistent airflow obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 40 and 80 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Confirmed diagnosis of COPD with forced expiratory volume in 1 second (FEV1) over forced vital capacity (FVC) ratio (FEV1/FVC) < 0.7, AND FEV1 < 80% and ≥ 30% predicted.
* Current or former smoker with a cigarette smoking history of ≥ 10 pack-years.
* Stable COPD patient with documented history of at least 1 moderate or severe acute exacerbation of COPD within the 12 months before Screening.
* Regular sputum producer.
* Capable to comply with the daily electronic Diary Card completion throughout the study period, according to investigator's judgement at Visit 1.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/ product.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine, with the exception of any influenza or pneumococcal vaccine which may be administered ≥ 15 days preceding or following any study vaccine dose.
* Previous vaccination with any vaccine containing NTHi antigens.
* Administration of immunoglobulins or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of non-steroid immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of immune-mediated disease other than COPD.
* Administration of systemic corticosteroids within the 30 days before Screening.
* Administration of systemic antibiotics within the 30 days before Screening.
* Chronic use of antibiotics for prevention of acute exacerbations of COPD (AECOPD).
* Receiving oxygen therapy.
* Planned lung transplantation.
* Planned/ underwent lung resection surgery.
* Diagnosis of α-1 antitrypsin deficiency as the underlying cause of COPD.
* Diagnosed with a respiratory disorder other than COPD, or chest X-ray/ CT scan revealing evidence of clinically significant abnormalities not believed to be due to the presence of COPD. Subjects with allergic rhinitis can be enrolled.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines and/ or the bronchodilator used for spirometry assessment during the study.
* Contraindication for spirometry testing.
* Clinically significant abnormality in haematology or biochemistry parameter.
* Acute cardiac insufficiency.
* Malignancies within the previous 5 years or lymphoproliferative disorder.
* Any known disease or condition likely to cause death during the study period.
* Acute disease and/ or fever at the time of Screening.

  * Fever is defined as oral or axillary temperature ≥ 37.5°C. The preferred route for recording temperature in this study will be oral.
  * Subjects with acute disease and/ or fever at the time of Screening may be enrolled at a later date if enrolment is still open. Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Current alcoholism and/or drug abuse.
* Other condition which the investigator judges may put the safety of the subject at risk through study participation or which may interfere with the study findings.
* Planned move to a location that will complicate participation in the trial through study end.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Örebro
- United Kingdom (11):
  - GSK Investigational Site, Llanelli, Carmarthenshire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Stoke-on-Trent, Staffordshire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Poole, Dorset
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Wolverhampton

REFERENCES:
- [Derived] Baffetta F, Buonsanti C, Moraschini L, Aprea S, Cane M, Lombardi S, Contorni M, Rondini S, Arora AK, Bardelli M, Finco O, Serruto D, Paccani SR. Lung mucosal immunity to NTHi vaccine antigens: Antibodies in sputum of chronic obstructive pulmonary disease patients. Hum Vaccin Immunother. 2024 Dec 31;20(1):2343544. doi: 10.1080/21645515.2024.2343544. Epub 2024 Apr 24. PMID 38655676
- [Derived] Wilkinson TMA, Schembri S, Brightling C, Bakerly ND, Lewis K, MacNee W, Rombo L, Hedner J, Allen M, Walker PP, De Ryck I, Tasciotti A, Casula D, Moris P, Testa M, Arora AK. Non-typeable Haemophilus influenzae protein vaccine in adults with COPD: A phase 2 clinical trial. Vaccine. 2019 Sep 24;37(41):6102-6111. doi: 10.1016/j.vaccine.2019.07.100. Epub 2019 Aug 22. PMID 31447126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 145 subjects, aged 40 to 80 years were recruited from 4 sites in Sweden and 11 sites in the United Kingdom.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- 10-AS01E Group: Approximately 70 subjects who received 2 doses of the investigational NTHi vaccine.
- Control Group: Approximately 70 subjects who received 2 doses of placebo.
Period: Overall Study
Arm/Group | 10-AS01E Group | Control Group
Started | 73 | 72
Completed | 69 | 64
Not Completed | 4 | 8
Not completed — Serious Adverse Event | 1 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Sponsor study termination | 0 | 1
Not completed — Other- unable to perform study procedure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10-AS01E Group | Control Group | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (8.41) | 66.8 (7.21) | 66.9 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 39 | 36 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White- Caucasian/ European Heritage | 73 | 72 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs).
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (from Day 0 to Day 6) after first dose.
Population: Analysis was performed on the Total Vaccinated Cohort (TVC) that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants
  Any Pain | 49 | 5
  Any Redness (mm) | 9 | 0
  Any Swelling (mm) | 4 | 0

2. Primary Outcome: Number of Subjects With Any Solicited Local AEs.
Description: as for outcome 1
Time Frame: During a 7-day follow-up period (from Day 60 to Day 66) after second dose.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 69 | 68
Participants
  Any Pain | 49 | 5
  Any Redness (mm) | 15 | 2
  Any Swelling (mm) | 8 | 0

3. Primary Outcome: Number of Subjects With Any Solicited General AEs.
Description: Assessed solicited general symptoms are fatigue, gastrointestinal symptoms (included nausea, vomiting, diarrhoea and/or abdominal pain), headache, fever [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (from Day 0 to Day 6) following the first dose.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants
  Any Fatigue | 21 | 19
  Any Gastrointestinal symptoms | 12 | 10
  Any Headache | 19 | 13
  Any Temperature/(Oral) (°C) | 2 | 6

4. Primary Outcome: Number of Subjects With Any Solicited General AEs
Description: Assessed solicited general symptoms are fatigue, gastrointestinal symptoms (included nausea, vomiting, diarrhoea and/or abdominal pain), headache, fever (defined as oral temperature equal to or above 37.5 °C). Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (from Day 60 to Day 66) following the second dose.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 69 | 68
Participants
  Any Fatigue | 28 | 13
  Any Gastrointestinal symptoms | 15 | 6
  Any Headache | 20 | 13
  Any Temperature/(Oral) (°C) | 10 | 1

5. Primary Outcome: Number of Subjects With Any Unsolicited AEs.
Description: Assessed unsolicited AEs covered any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day follow-up period (from Day 0 to Day 29) following the first dose.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants | 27 | 26

6. Primary Outcome: Number of Subjects With Any Unsolicited AEs
Description: as for outcome 5
Time Frame: During the 30-day follow-up period (from Day 60 to Day 89) following the second dose.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants | 25 | 22

7. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: Assessed haematological parameters are complete blood cell count: Leukocytes [white blood cells (WBC)], differential count (basophils, eosinophils, lymphocytes, monocytes, neutrophils), platelets count, and hemoglobin level below or above the normal laboratory ranges tabulated by time point. Assessed biochemical parameters are alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatinine below or above the normal laboratory ranges tabulated by time point.
Time Frame: At Day 0.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 70
Participants
  WBC below: number analyzed (Participants) | 72 | 70
  WBC below | 1 | 1
  WBC above: number analyzed (Participants) | 72 | 70
  WBC above | 5 | 1
  Basophils below: number analyzed (Participants) | 71 | 70
  Basophils below | 0 | 0
  Basophils above: number analyzed (Participants) | 71 | 70
  Basophils above | 0 | 0
  Eosinophils below: number analyzed (Participants) | 71 | 70
  Eosinophils below | 0 | 0
  Eosinophils above: number analyzed (Participants) | 71 | 70
  Eosinophils above | 3 | 4
  Lymphocytes below: number analyzed (Participants) | 71 | 70
  Lymphocytes below | 15 | 9
  Lymphocytes above: number analyzed (Participants) | 71 | 70
  Lymphocytes above | 7 | 3
  Monocytes below: number analyzed (Participants) | 71 | 70
  Monocytes below | 0 | 1
  Monocytes above: number analyzed (Participants) | 71 | 70
  Monocytes above | 6 | 6
  Neutrophils below: number analyzed (Participants) | 71 | 70
  Neutrophils below | 1 | 1
  Neutrophils above: number analyzed (Participants) | 71 | 70
  Neutrophils above | 6 | 3
  Platelets below: number analyzed (Participants) | 72 | 70
  Platelets below | 2 | 4
  Platelets above: number analyzed (Participants) | 72 | 70
  Platelets above | 12 | 9
  Haemoglobin below: number analyzed (Participants) | 72 | 70
  Haemoglobin below | 5 | 6
  Haemoglobin above: number analyzed (Participants) | 72 | 70
  Haemoglobin above | 12 | 5
  ALT below: number analyzed (Participants) | 72 | 70
  ALT below | 0 | 0
  ALT above: number analyzed (Participants) | 72 | 70
  ALT above | 4 | 1
  AST below: number analyzed (Participants) | 72 | 70
  AST below | 0 | 0
  AST above: number analyzed (Participants) | 72 | 70
  AST above | 2 | 1
  Creatinine below | 0 | 0
  Creatinine above | 10 | 8

8. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 7.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 69 | 67
Participants
  WBC below | 0 | 2
  WBC above | 4 | 0
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 4 | 2
  Lymphocytes below | 9 | 7
  Lymphocytes above | 4 | 2
  Monocytes below | 1 | 0
  Monocytes above | 4 | 5
  Neutrophils below | 1 | 1
  Neutrophils above | 8 | 1
  Platelets below | 2 | 3
  Platelets above | 15 | 12
  Haemoglobin below | 5 | 5
  Haemoglobin above | 12 | 4
  ALT below | 0 | 0
  ALT above | 5 | 1
  AST below | 0 | 0
  AST above | 1 | 2
  Creatinine below | 0 | 0
  Creatinine above | 7 | 10

9. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 30.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 68 | 68
Participants
  WBC below | 1 | 1
  WBC above | 8 | 2
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 3 | 2
  Lymphocytes below | 14 | 6
  Lymphocytes above | 7 | 6
  Monocytes below | 0 | 0
  Monocytes above | 8 | 10
  Neutrophils below | 1 | 2
  Neutrophils above | 9 | 1
  Platelets below | 3 | 2
  Platelets above | 14 | 11
  Haemoglobin below | 3 | 8
  Haemoglobin above | 10 | 6
  ALT below | 0 | 0
  ALT above | 5 | 4
  AST below | 0 | 0
  AST above | 1 | 4
  Creatinine below | 0 | 0
  Creatinine above | 6 | 12

10. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 60.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 70 | 69
Participants
  WBC below | 1 | 0
  WBC above | 3 | 8
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 5 | 2
  Lymphocytes below | 12 | 11
  Lymphocytes above | 4 | 5
  Monocytes below | 0 | 2
  Monocytes above | 7 | 12
  Neutrophils below | 1 | 2
  Neutrophils above | 8 | 7
  Platelets below | 1 | 3
  Platelets above | 13 | 9
  Haemoglobin below | 4 | 8
  Haemoglobin above | 7 | 5
  ALT below: number analyzed (Participants) | 70 | 68
  ALT below | 0 | 0
  ALT above: number analyzed (Participants) | 70 | 68
  ALT above | 4 | 1
  AST below | 0 | 0
  AST above | 3 | 2
  Creatinine below | 0 | 0
  Creatinine above | 5 | 8

11. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 67.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 65 | 64
Participants
  WBC below | 0 | 0
  WBC above | 4 | 2
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 5 | 2
  Lymphocytes below | 11 | 8
  Lymphocytes above | 6 | 3
  Monocytes below | 0 | 0
  Monocytes above | 4 | 12
  Neutrophils below | 2 | 1
  Neutrophils above | 5 | 4
  Platelets below | 0 | 4
  Platelets above | 16 | 11
  Haemoglobin below | 6 | 11
  Haemoglobin above | 8 | 3
  ALT below: number analyzed (Participants) | 64 | 64
  ALT below | 0 | 0
  ALT above: number analyzed (Participants) | 64 | 64
  ALT above | 5 | 2
  AST below: number analyzed (Participants) | 64 | 64
  AST below | 0 | 0
  AST above: number analyzed (Participants) | 64 | 64
  AST above | 3 | 3
  Creatinine below: number analyzed (Participants) | 64 | 64
  Creatinine below | 0 | 0
  Creatinine above: number analyzed (Participants) | 64 | 64
  Creatinine above | 5 | 9

12. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 90.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 72 | 69
Participants
  WBC below | 0 | 1
  WBC above | 3 | 2
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 7 | 5
  Lymphocytes below | 11 | 10
  Lymphocytes above | 6 | 4
  Monocytes below | 0 | 0
  Monocytes above | 10 | 6
  Neutrophils below | 1 | 0
  Neutrophils above | 5 | 5
  Platelets below | 1 | 3
  Platelets above | 13 | 13
  Haemoglobin below | 4 | 10
  Haemoglobin above | 10 | 6
  ALT below | 0 | 0
  ALT above | 3 | 4
  AST below | 0 | 0
  AST above | 2 | 2
  Creatinine below | 0 | 0
  Creatinine above | 5 | 8

13. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 270.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 67 | 65
Participants
  WBC below | 1 | 0
  WBC above | 7 | 5
  Basophils below | 0 | 0
  Basophils above | 0 | 0
  Eosinophils below | 0 | 0
  Eosinophils above | 4 | 3
  Lymphocytes below | 11 | 5
  Lymphocytes above | 7 | 3
  Monocytes below | 0 | 0
  Monocytes above | 10 | 9
  Neutrophils below | 1 | 1
  Neutrophils above | 10 | 6
  Platelets below | 1 | 3
  Platelets above | 9 | 11
  Haemoglobin below | 5 | 10
  Haemoglobin above | 13 | 3
  ALT below | 0 | 0
  ALT above | 5 | 2
  AST below | 0 | 0
  AST above | 5 | 2
  Creatinine below | 0 | 0
  Creatinine above | 9 | 9

14. Primary Outcome: Number of Subjects With Each Haematological/ Biochemical Laboratory Abnormality.
Description: as for outcome 7
Time Frame: At Day 450.
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 69 | 61
Participants
  WBC below: number analyzed (Participants) | 68 | 61
  WBC below | 1 | 0
  WBC above: number analyzed (Participants) | 68 | 61
  WBC above | 3 | 1
  Basophils below: number analyzed (Participants) | 68 | 60
  Basophils below | 0 | 0
  Basophils above: number analyzed (Participants) | 68 | 60
  Basophils above | 0 | 0
  Eosinophils below: number analyzed (Participants) | 68 | 60
  Eosinophils below | 0 | 0
  Eosinophils above: number analyzed (Participants) | 68 | 60
  Eosinophils above | 6 | 3
  Lymphocytes below: number analyzed (Participants) | 68 | 60
  Lymphocytes below | 17 | 9
  Lymphocytes above: number analyzed (Participants) | 68 | 60
  Lymphocytes above | 8 | 3
  Monocytes below: number analyzed (Participants) | 68 | 60
  Monocytes below | 0 | 1
  Monocytes above: number analyzed (Participants) | 68 | 60
  Monocytes above | 6 | 5
  Neutrophils below: number analyzed (Participants) | 68 | 60
  Neutrophils below | 1 | 1
  Neutrophils above: number analyzed (Participants) | 68 | 60
  Neutrophils above | 7 | 4
  Platelets below: number analyzed (Participants) | 68 | 61
  Platelets below | 3 | 3
  Platelets above: number analyzed (Participants) | 68 | 61
  Platelets above | 14 | 13
  Haemoglobin below: number analyzed (Participants) | 68 | 61
  Haemoglobin below | 6 | 10
  Haemoglobin above: number analyzed (Participants) | 68 | 61
  Haemoglobin above | 10 | 6
  ALT below | 0 | 0
  ALT above | 3 | 3
  AST below | 0 | 0
  AST above | 1 | 3
  Creatinine below | 0 | 0
  Creatinine above | 7 | 9

15. Primary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs).
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination (Day 0) up to study conclusion (Day 450).
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants | 2 | 0

16. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity or are a congenital anomaly/ birth defect in the offspring of a study subject.
Time Frame: From first vaccination (Day 0) up to study conclusion (Day 450).
Population: Analysis was performed on the TVC that included all subjects with at least 1 study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 73 | 72
Participants | 15 | 17

17. Secondary Outcome: Concentration of Anti Protein D (Anti-PD) Total Immunoglobulin G (IgG) Antibodies Against the NTHi Vaccine Antigens.
Description: Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay was 153 EL.U/mL for anti-PD.
Time Frame: At Day 0, Day 30, Day 60, Day 90, Day 270 and at Day 450.
Population: Analysis was performed on the According to Protocol (ATP) cohort for Immunogenicity which included all evaluable subjects who received the study vaccine according to their treatment assigned and for whom post-vaccination immunogenicity results were available for at least 1 assay.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 46 | 45
EL.U/mL
  Anti-PD antibody, Day 0: number analyzed (Participants) | 44 | 45
  Anti-PD antibody, Day 0 | 107.3 [87.9 to 130.9] | 100.3 [85.3 to 118]
  Anti-PD antibody, Day 30: number analyzed (Participants) | 43 | 44
  Anti-PD antibody, Day 30 | 840.1 [535.9 to 1317] | 102.6 [86.2 to 122.1]
  Anti-PD antibody, Day 60 | 538 [358.6 to 807.1] | 104.1 [87.6 to 123.6]
  Anti-PD antibody, Day 90 | 1692.1 [1242.6 to 2304] | 103 [87.3 to 121.7]
  Anti-PD antibody, Day 270: number analyzed (Participants) | 44 | 42
  Anti-PD antibody, Day 270 | 598.3 [437 to 819.2] | 109.3 [90.9 to 131.4]
  Anti-PD antibody, Day 450: number analyzed (Participants) | 46 | 41
  Anti-PD antibody, Day 450 | 463 [340.4 to 629.8] | 108.4 [90.1 to 130.4]

18. Secondary Outcome: Concentration of Anti Protein E (Anti-PE) Total IgG Antibodies Against the NTHi Vaccine Antigens.
Description: Antibody concentrations were measured by ELISA and expressed as GMCs in EL.U/mL. The cut-off of the assay was 8 EL.U/mL for anti-PE.
Time Frame: At Day 0, Day 30, Day 60, Day 90, Day 270 and at Day 450
Population: Analysis was performed on the ATP cohort for Immunogenicity which included all evaluable subjects who received the study vaccine according to their treatment assigned and for whom post-vaccination immunogenicity results were available for at least 1 assay.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 46 | 44
EL.U/mL
  Anti-PE antobody, Day 0: number analyzed (Participants) | 43 | 44
  Anti-PE antobody, Day 0 | 14.1 [9.5 to 21] | 14.8 [10.2 to 21.5]
  Anti-PE antobody, Day 30: number analyzed (Participants) | 43 | 43
  Anti-PE antobody, Day 30 | 1007 [588.9 to 1722] | 13.6 [9.4 to 19.5]
  Anti-PE antobody, Day 60 | 823.7 [503.3 to 1348.1] | 13.9 [9.7 to 19.9]
  Anti-PE antobody, Day 90: number analyzed (Participants) | 44 | 44
  Anti-PE antobody, Day 90 | 10953.4 [8414.9 to 14257.9] | 15 [10.3 to 21.9]
  Anti-PE antobody, Day 270: number analyzed (Participants) | 44 | 41
  Anti-PE antobody, Day 270 | 1743.3 [1226.9 to 2477] | 12.6 [8.7 to 18.1]
  Anti-PE antobody, Day 450: number analyzed (Participants) | 46 | 40
  Anti-PE antobody, Day 450 | 1247.5 [866 to 1797] | 13.6 [9.3 to 20]

19. Secondary Outcome: Concentration of Anti-PilA Total IgG Antibodies Against the NTHi Vaccine Antigens.
Description: Antibody concentrations were measured by ELISA and expressed as GMCs in EL.U/mL. The cut-off of the assay was 7 EL.U/mL for anti-PilA.
Time Frame: At Day 0, Day 30, Day 60, Day 90, Day 270 and at Day 450.
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: El.U/mL
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 46 | 43
El.U/mL
  Anti-PilA antibody, Day 0: number analyzed (Participants) | 39 | 43
  Anti-PilA antibody, Day 0 | 12.3 [8.6 to 17.6] | 14.5 [10.2 to 20.5]
  Anti-PilA antibody, Day 30: number analyzed (Participants) | 41 | 40
  Anti-PilA antibody, Day 30 | 234.3 [133.5 to 411.5] | 15.6 [10.7 to 22.8]
  Anti-PilA antibody, Day 60: number analyzed (Participants) | 43 | 43
  Anti-PilA antibody, Day 60 | 207.5 [122.4 to 351.6] | 15.1 [10.7 to 21.3]
  Anti-PilA antibody, Day 90: number analyzed (Participants) | 46 | 41
  Anti-PilA antibody, Day 90 | 1353.7 [989.7 to 1851.7] | 16.5 [11.4 to 23.9]
  Anti-PilA antibody, Day 270: number analyzed (Participants) | 43 | 39
  Anti-PilA antibody, Day 270 | 333.5 [240.2 to 463.2] | 16.8 [11.6 to 24.3]
  Anti-PilA antibody, Day 450: number analyzed (Participants) | 45 | 38
  Anti-PilA antibody, Day 450 | 206.8 [147.7 to 289.5] | 16.2 [11.1 to 23.6]

20. Secondary Outcome: Frequency of Specific Cluster of Differentiation 4 (CD4+) T-cells Against NTHi Antigens Collected for Evaluation of Cell-mediated Immune Response.
Description: Frequency of specific CD4+ T-cells were measured by flow cytometry intracellular cytokine staining (ICS) expressing two or more markers [such as Interleukin-2 (IL-2), IL-13, IL-17, Interferon-γ (IFN-γ), Tumor Necrosis Factor-α (TNF-α) and Cluster of Differentiation 40 Ligand (CD40L)].The frequency of specific CD4+ T-cells are summarised [descriptive statistics: Mean and standard deviation (SD)] against each antigen (PD, PE and PilA), by group at each time point during which blood samples are collected for CMI.
Time Frame: At Day 0, Day 90, Day 270 and at Day 450.
Population: Analysis was performed on a sub-cohort of participants from the ATP cohort for Immunogenicity, including approximately 40 subjects (20/each group), for which an additional blood sample was taken at the specified time points. The analysis was only performed on those subjects with available results for the analyzed outcome variable.
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/ million cells
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 15 | 9
CD4+ T-cells/ million cells
  CD4+ T-cells, PD, Day 0: number analyzed (Participants) | 15 | 7
  CD4+ T-cells, PD, Day 0 | 33.1 (49.97) | 79.7 (91.48)
  CD4+ T-cells, PD, Day 90: number analyzed (Participants) | 15 | 8
  CD4+ T-cells, PD, Day 90 | 521.6 (287.39) | 38.4 (51.61)
  CD4+ T-cells, PD, Day 270: number analyzed (Participants) | 14 | 9
  CD4+ T-cells, PD, Day 270 | 189.6 (146.87) | 51.8 (59.4)
  CD4+ T-cells, PD, Day 450: number analyzed (Participants) | 14 | 5
  CD4+ T-cells, PD, Day 450 | 148.6 (141.11) | 97.8 (98.4)
  CD4+ T-cells, PE, Day 0: number analyzed (Participants) | 15 | 8
  CD4+ T-cells, PE, Day 0 | 51.3 (68.72) | 69.1 (82.87)
  CD4+ T-cells, PE, Day 90: number analyzed (Participants) | 15 | 8
  CD4+ T-cells, PE, Day 90 | 857.9 (642.76) | 65 (92.86)
  CD4+ T-cells, PE, Day 270: number analyzed (Participants) | 14 | 9
  CD4+ T-cells, PE, Day 270 | 304.4 (292.46) | 71.6 (90.51)
  CD4+ T-cells, PE, Day 450: number analyzed (Participants) | 14 | 5
  CD4+ T-cells, PE, Day 450 | 337.2 (302.42) | 117.8 (53.24)
  CD4+ T-cells, PilA, Day 0: number analyzed (Participants) | 15 | 7
  CD4+ T-cells, PilA, Day 0 | 29.7 (53.21) | 98.3 (74.27)
  CD4+ T-cells, PilA, Day 90: number analyzed (Participants) | 15 | 8
  CD4+ T-cells, PilA, Day 90 | 474.4 (321.58) | 37.4 (46.53)
  CD4+ T-cells, PilA, Day 270: number analyzed (Participants) | 14 | 9
  CD4+ T-cells, PilA, Day 270 | 145 (164.58) | 80.3 (95.6)
  CD4+ T-cells, PilA, Day 450: number analyzed (Participants) | 14 | 5
  CD4+ T-cells, PilA, Day 450 | 157.7 (117.76) | 102.8 (116.48)

21. Secondary Outcome: Frequency of Specific CD8+ T-cells Against NTHi Antigens Collected for Evaluation of Cell-mediated Immune Response.
Description: Frequency of specific CD8+ T-cells were measured by flow cytometry ICS expressing two or more markers (such as IL-2, IL-13, IL-17, IFN-γ, TNF-α and CD40L).The frequency of specific CD8+ T-cells are summarised [descriptive statistics: Mean and standard deviation (SD)] against each antigen (PD, PE and PilA), by group at each time point during which blood samples are collected for CMI.
Time Frame: At Day 0, Day 90, Day 270 and at Day 450.
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: CD8+ T-cells/ million cells
Arm/Group | 10-AS01E Group | Control Group
Number analyzed (Participants) | 14 | 9
CD8+ T-cells/ million cells
  CD8+ T-cells, PD, Day 0: number analyzed (Participants) | 13 | 8
  CD8+ T-cells, PD, Day 0 | 97.1 (186.24) | 47.9 (72.9)
  CD8+ T-cells, PD, Day 90: number analyzed (Participants) | 12 | 8
  CD8+ T-cells, PD, Day 90 | 39.6 (73.78) | 45.8 (77.53)
  CD8+ T-cells, PD, Day 270: number analyzed (Participants) | 12 | 9
  CD8+ T-cells, PD, Day 270 | 55.3 (59.18) | 48.7 (56.33)
  CD8+ T-cells, PD, Day 450: number analyzed (Participants) | 13 | 5
  CD8+ T-cells, PD, Day 450 | 51.5 (60.19) | 16.2 (24.04)
  CD8+ T-cells, PE, Day 0: number analyzed (Participants) | 14 | 8
  CD8+ T-cells, PE, Day 0 | 97.7 (204.06) | 73.9 (131.71)
  CD8+ T-cells, PE, Day 90: number analyzed (Participants) | 14 | 8
  CD8+ T-cells, PE, Day 90 | 44.9 (47.72) | 30.6 (59.01)
  CD8+ T-cells, PE, Day 270: number analyzed (Participants) | 12 | 9
  CD8+ T-cells, PE, Day 270 | 29.9 (57.16) | 60.3 (83.47)
  CD8+ T-cells, PE, Day 450: number analyzed (Participants) | 13 | 5
  CD8+ T-cells, PE, Day 450 | 41 (74.41) | 31.6 (43.34)
  CD8+ T-cells, PilA, Day 0: number analyzed (Participants) | 13 | 8
  CD8+ T-cells, PilA, Day 0 | 63.1 (122.12) | 23.1 (45.92)
  CD8+ T-cells, PilA, Day 90: number analyzed (Participants) | 13 | 8
  CD8+ T-cells, PilA, Day 90 | 39.7 (73.42) | 80.3 (125.84)
  CD8+ T-cells, PilA, Day 270: number analyzed (Participants) | 12 | 9
  CD8+ T-cells, PilA, Day 270 | 27.4 (34.15) | 13 (15.12)
  CD8+ T-cells, PilA, Day 450: number analyzed (Participants) | 13 | 5
  CD8+ T-cells, PilA, Day 450 | 63.7 (98.87) | 31 (36.17)

ADVERSE EVENTS:
Time Frame: Solicted AEs: during the 7-day interval post each vaccine dose, Unsolicited AEs: during the 30-day interval post each vaccine dose, SAEs: throughout the entire study, from Day 0 up to Day 450.
Arm/Group | 10-AS01E Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/73 | 2/72
Serious Adverse Events (participants affected / at risk) | 15/73 | 17/72
Other Adverse Events (participants affected / at risk) | 65/73 | 42/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10-AS01E Group (N=73) | Control Group (N=72)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (3) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 10 (14)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10-AS01E Group (N=73) | Control Group (N=72)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 37 (51) | 23 (32)
Gastrointestinal disorder (Gastrointestinal disorders) | 22 (27) | 15 (16)
Headache (Nervous system disorders) | 30 (42) | 22 (34)
Injection site erythema (General disorders) | 19 (26) | 2 (2)
Injection site pain (General disorders) | 59 (98) | 9 (10)
Injection site swelling (General disorders) | 9 (12) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Pyrexia (General disorders) | 10 (12) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT02075541/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT02075541/SAP_001.pdf